CLINICAL TRIAL: NCT06120088
Title: U.S Guided Erector Spinae Block for Postoperative Pain Control in Patients Undergoing Para Umblical Hernial Repair. (Comparative Study ).
Brief Title: U.S. Guided Erector Spinae Block for Postoperative Pain Management in Paraumbilical Hernia Repair Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Ahmed Hussien, Dr, Assiut University
Other Study IDs: US-ESB for Postop Pain Control
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Regional Anesthesia
MeSH Terms: interventions — Dexamethasone; Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The Bupivacaine: Patients in this group received bilateral ultrasound-guided erector spinae plane block at the level of T7 transverse process using 20 mL of bupivacaine 0.25% on each side + 1ml saline placebo.
  Interventions: Drug: Bubpivacaine
- The Bubpivacaine and dexamethasone: Patients in this group received bilateral ultrasound-guided erector spinae plane block at the level of T7 transverse process using 20 mL of bupivacaine 0.25% plus 1ml dexamethasone on each side
  Interventions: Drug: Bubpivacaine; Drug: dexamethasone
- The Bubpivacaine and fentanyl: Patients in this group received bilateral ultrasound-guided erector spinae plane block at the level of T7 transverse process using 20 mL of bupivacaine 0.25% in addition to calculated dose of fentanyl on each side
  Interventions: Drug: Bubpivacaine; Drug: fentanyl

INTERVENTIONS:
Drug: Bubpivacaine — Bupivacaine is a long-acting local anesthetic commonly used to provide pain relief by blocking nerve signals in a specific area. It's often utilized for various medical procedures and surgeries, offering prolonged numbing effects.
Drug: dexamethasone — Dexamethasone is a potent corticosteroid with anti-inflammatory properties. It's frequently employed as an adjunct in medical treatments to reduce inflammation and swelling, and in some cases, to prevent nausea and vomiting associated with certain medications or procedures.
  Groups: The Bubpivacaine and dexamethasone
Drug: fentanyl — Fentanyl is a powerful synthetic opioid pain reliever. It acts on the central nervous system to alleviate severe pain. Fentanyl is significantly potent and is used in medical settings for acute pain management, such as during surgeries or for chronic pain in cases where other opioids may not be as effective.
  Groups: The Bubpivacaine and fentanyl

SUMMARY:
Abdominal surgery is one of the most definitive and mainstay treatment options for abdominal pathologies in clinical practice. Acute postoperative pain is a major challenge in the postoperative period. Although opioids are commonly used for analgesia after paraumbilical hernia, they can lead to side effects, such as nausea and vomiting, constipation, pruritus, and life-threatening respiratory depression. Regional anesthetic techniques are commonly used to prevent or minimize these side effects. The objective of this study is to assess the effectiveness of erector spinae plane block (ESPB) and standard medical (no block) pain management after paraumbilical hernia.

ELIGIBILITY:
Inclusion Criteria:

* Age group : 18-60 years old
* Both genders
* Patient scheduled for paraumbilical hernia surgeries

Exclusion Criteria:

* Allergy to medications used in this study
* Patient's refusal to participate in this study
* Recurrent cases
* Any complications to local blocks
* Emergency surgical procedures

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Sample size was calculated using G power 3.1.9.2. To be able to calculate the difference in first analgesic request between the three studied groups with α error of 0.05, power of study of 0.9, equal group assignment and 0.4 effect size and using ANOVA test for comparison we need to include 27 patients in each group, another 3 patients will be added to each group to compensate for violation at the study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
first analgesic request | baseline
  signifies the initial instance when a patient asks for pain relief, commonly occurring post-surgery or during medical care, marking the first acknowledgment or complaint of discomfort prompting the need for pain medication or management.

SECONDARY OUTCOMES:
VAS score | baseline
  a quantitative measure used in healthcare to assess and quantify pain levels. It involves a patient marking their perceived pain intensity on a 10-point or 100-point scale, typically from "no pain" to "worst pain imaginable," providing a straightforward and subjective representation of pain severity.

REFERENCES:
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Ohkura Y, Shindoh J, Ueno M, Iizuka T, Haruta S, Udagawa H. A new postoperative pain management (intravenous acetaminophen: Acelio(R)) leads to enhanced recovery after esophagectomy: a propensity score-matched analysis. Surg Today. 2018 May;48(5):502-509. doi: 10.1007/s00595-017-1616-5. Epub 2017 Dec 12. PMID 29234960
- [Background] Crumley S, Schraag S. The role of local anaesthetic techniques in ERAS protocols for thoracic surgery. J Thorac Dis. 2018 Mar;10(3):1998-2004. doi: 10.21037/jtd.2018.02.48. PMID 29707356
- [Background] Boisen ML, Sardesai MP, Kolarczyk L, Rao VK, Owsiak CP, Gelzinis TA. The Year in Thoracic Anesthesia: Selected Highlights From 2017. J Cardiothorac Vasc Anesth. 2018 Aug;32(4):1556-1569. doi: 10.1053/j.jvca.2018.03.001. Epub 2018 Mar 13. No abstract available. PMID 29655515
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Viderman D, Dautova A, Sarria-Santamera A. Erector spinae plane block in acute interventional pain management: a systematic review. Scand J Pain. 2021 May 14;21(4):671-679. doi: 10.1515/sjpain-2020-0171. Print 2021 Oct 26. PMID 33984888
- [Background] Viderman D, Sarria-Santamera A. Erector spinae plane block in chronic pain management: a scoping review. Tumori. 2021 Oct;107(5):458-467. doi: 10.1177/0300891620985935. Epub 2021 Jan 12. PMID 33430714
- [Background] Luo D, Wan X, Liu J, Tong T. Optimally estimating the sample mean from the sample size, median, mid-range, and/or mid-quartile range. Stat Methods Med Res. 2018 Jun;27(6):1785-1805. doi: 10.1177/0962280216669183. Epub 2016 Sep 27. PMID 27683581
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443
- [Background] Knotkova H, Fine PG, Portenoy RK. Opioid rotation: the science and the limitations of the equianalgesic dose table. J Pain Symptom Manage. 2009 Sep;38(3):426-39. doi: 10.1016/j.jpainsymman.2009.06.001. PMID 19735903
- [Background] Mercadante S, Caraceni A. Conversion ratios for opioid switching in the treatment of cancer pain: a systematic review. Palliat Med. 2011 Jul;25(5):504-15. doi: 10.1177/0269216311406577. PMID 21708857
- [Background] Santonocito C, Noto A, Crimi C, Sanfilippo F. Remifentanil-induced postoperative hyperalgesia: current perspectives on mechanisms and therapeutic strategies. Local Reg Anesth. 2018 Apr 9;11:15-23. doi: 10.2147/LRA.S143618. eCollection 2018. PMID 29670398
- [Background] Abdelhamid BM, Khaled D, Mansour MA, Hassan MM. Comparison between the ultrasound-guided erector spinae block and the subcostal approach to the transversus abdominis plane block in obese patients undergoing sleeve gastrectomy: a randomized controlled trial. Minerva Anestesiol. 2020 Aug;86(8):816-826. doi: 10.23736/S0375-9393.20.14064-1. Epub 2020 May 22. PMID 32449336
- [Background] Abu Elyazed MM, Mostafa SF, Abdelghany MS, Eid GM. Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Open Epigastric Hernia Repair: A Prospective Randomized Controlled Study. Anesth Analg. 2019 Jul;129(1):235-240. doi: 10.1213/ANE.0000000000004071. PMID 30801359
- [Background] Hamed MA, Goda AS, Basiony MM, Fargaly OS, Abdelhady MA. Erector spinae plane block for postoperative analgesia in patients undergoing total abdominal hysterectomy: a randomized controlled study original study. J Pain Res. 2019 Apr 30;12:1393-1398. doi: 10.2147/JPR.S196501. eCollection 2019. PMID 31118757
- [Background] Kamel AAF, Amin OAI, Ibrahem MAM. Bilateral Ultrasound-Guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block on Postoperative Analgesia after Total Abdominal Hysterectomy. Pain Physician. 2020 Jul;23(4):375-382. PMID 32709172
- [Background] Kim D, Kim JM, Choi GS, Heo G, Kim GS, Jeong JS. Ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic liver resection: A prospective, randomised controlled, patient and observer-blinded study. Eur J Anaesthesiol. 2021 Aug 1;38(Suppl 2):S106-S112. doi: 10.1097/EJA.0000000000001475. PMID 33653982
- [Background] Prasad MK, Varshney RK, Jain P, Choudhary AK, Khare A, Jheetay GS. Postoperative analgesic efficacy of fluoroscopy-guided erector spinae plane block after percutaneous nephrolithotomy (PCNL): A randomized controlled study. Saudi J Anaesth. 2020 Oct-Dec;14(4):480-486. doi: 10.4103/sja.SJA_26_20. Epub 2020 Sep 24. PMID 33447190
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Zhang Y, Liu T, Zhou Y, Yu Y, Chen G. Analgesic efficacy and safety of erector spinae plane block in breast cancer surgery: a systematic review and meta-analysis. BMC Anesthesiol. 2021 Feb 20;21(1):59. doi: 10.1186/s12871-021-01277-x. PMID 33610172
- [Background] Wigmore T, Farquhar-Smith P. Opioids and cancer: friend or foe? Curr Opin Support Palliat Care. 2016 Jun;10(2):109-18. doi: 10.1097/SPC.0000000000000208. PMID 26990052
- [Background] Hickey OT, Burke SM, Hafeez P, Mudrakouski AL, Hayes ID, Shorten GD. Severity of acute pain after breast surgery is associated with the likelihood of subsequently developing persistent pain. Clin J Pain. 2010 Sep;26(7):556-60. doi: 10.1097/AJP.0b013e3181dee988. PMID 20639740
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Kuscu Y, Gumus Demirbilek S. Ultrasound-guided erector spinae plane block versus oblique subcostal transversus abdominis plane block for postoperative analgesia of adult patients undergoing laparoscopic cholecystectomy: Randomized, controlled trial. J Clin Anesth. 2019 Nov;57:31-36. doi: 10.1016/j.jclinane.2019.03.012. Epub 2019 Mar 6. PMID 30851501
- [Background] Temirov T, Ben-David B, Mustafin A, Viderman D. Erector Spinae Plane Block in Management of Pain After Kidney Transplantation. Pain Med. 2019 May 1;20(5):1053-1054. doi: 10.1093/pm/pny221. No abstract available. PMID 30412258
- [Background] Chin KJ, Chan V. Ultrasound-guided peripheral nerve blockade. Curr Opin Anaesthesiol. 2008 Oct;21(5):624-31. doi: 10.1097/ACO.0b013e32830815d1. PMID 18784490
- [Background] Viderman D, Ben-David B, Sarria-Santamera A. Analysis of bupivacaine and ropivacaine-related cardiac arrests in regional anesthesia: A systematic review of case reports. Rev Esp Anestesiol Reanim (Engl Ed). 2021 Oct;68(8):472-483. doi: 10.1016/j.redare.2020.10.005. Epub 2021 Sep 17. PMID 34538765
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Gumus Demirbilek S. Comparison of the efficacy of erector spinae plane block performed with different concentrations of bupivacaine on postoperative analgesia after mastectomy surgery: ramdomized, prospective, double blinded trial. BMC Anesthesiol. 2019 Mar 4;19(1):31. doi: 10.1186/s12871-019-0700-3. PMID 30832580